CLINICAL TRIAL: NCT02231918
Title: An Open-label Clinical Study to Investigate Pharmacokinetics (PK) of Different Doses (0.125 mg, 0.25 mg, 0.5 mg) of Pramipexole Administered Once Daily Orally in Pediatric Patients Who Are Individually Optimized to Stable Pramipexole Doses for the Treatment of Idiopathic Restless Legs Syndrome (RLS)
Brief Title: Study to Investigate Pharmacokinetics (PK) of Pramipexole in Pediatric Patients Who Are Individually Optimized to Stable Pramipexole Doses for the Treatment of Idiopathic Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 248.600
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

ARMS (3):
- MIRAPEX® - low (Experimental)
  Interventions: Drug: MIRAPEX® - low
- MIRAPEX® - medium (Experimental)
  Interventions: Drug: MIRAPEX® - medium
- MIRAPEX® - high (Experimental)
  Interventions: Drug: MIRAPEX® - high

INTERVENTIONS:
Drug: MIRAPEX® - low
  Arms: MIRAPEX® - low
Drug: MIRAPEX® - medium
  Arms: MIRAPEX® - medium
Drug: MIRAPEX® - high
  Arms: MIRAPEX® - high

SUMMARY:
Study to determine the pharmacokinetics (PK) of pramipexole (PPX) after administration of a single dose orally (p.o.) in pediatric patients with the diagnosis of RLS

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages 6 years to 16 years (two age groups, 6 to 11 years and 12 to 16 years, with the same number of patients if possible)
2. Diagnosis of idiopathic Restless Legs Syndrome (RLS) according to the Clinical RLS criteria of the International Restless Legs Syndrome Study Group (IRLSSG)

   All 4 of the following criteria must be present:
   * An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs. (Sometimes the urge to move is present without the uncomfortable sensations and sometimes the arms or other body parts are involved in addition to the legs.)
   * The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting
   * The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues
   * The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night. (When symptoms are very severe, the worsening at night may not be noticeable but must have been previously present.)
3. Must meet all 4 of the diagnostic criteria for adult RLS (see inclusion criterion No. 2 above) and either:

   1. The child must be able to describe the leg discomfort in their own words or
   2. The child must have 2 or 3 of the following:

      * Sleep disturbance
      * Periodic Limb Movements During Sleep (PLMS) index >5 per hour of sleep, or
      * A biological parent or sibling with definite RLS
4. Written informed consent consistent with International Conference on Harmonisation (ICH)/ Good Clinical Practice (GCP) and Local Institutional Review Board requirements for children obtained prior to any study procedures being performed
5. Ability and willingness to comply with the study treatment regimen and to attend study assessments
6. Must be on PPX treatment at the same evening maintenance dose for a minimum of 7 days prior to entry into this study as determined by the investigator
7. A patient who is taking PPX but not as an evening maintenance dose may return for a repeat screening if the patient can be successfully switched and re-stabilized to an evening PPX maintenance dose

Exclusion criteria:

1. Any women of childbearing potential having a positive serum pregnancy test at screening
2. Any women of childbearing potential not using a medically accepted method of contraceptive (Intra-Uterine Device, oral, implantable, injectable contraceptives and estrogen patch, double barrier method [spermicide + diaphragm], or abstinence at the discretion of the investigator)
3. Patients who have a clinically significant renal disease or serum creatinine level greater than 1.0 mg/dL at screening
4. Any of the following lab results at screening:

   * Hemoglobin (Hgb) below the lower limit of normal (LLN), which is determined to be clinically significant
   * Basal thyroid stimulating hormone (TSH), triiodothyronine (T3) or thyroxine (T4) clinically significantly (at the investigator's discretion) out of the normal range at screening (if not caused by substitution therapy according to the investigator's opinion)
   * Patients with any clinically significant abnormalities in laboratory parameters at screening at the investigator's discretion
5. Other clinically significant metabolic-endocrine, hematological, gastrointestinal disease, pulmonary disease (such as severe asthma) which in the opinion of the investigator would preclude the patient from participating in this study
6. History or clinical signs of any neurological disease with potential to secondarily cause RLS symptoms
7. Presence of any other sleep disorder such as Rapid Eye Movement (REM) sleep behavior disorder, narcolepsy, or sleep apnea syndrome
8. History of schizophrenia or any psychotic disorder, history of mental disorders, or any present Axis I psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) requiring any medical therapy
9. History of/or clinical signs of epilepsy or seizures other than fever-related seizures in early childhood
10. History of/or clinical signs of any malignant neoplasm including suspicious undiagnosed skin lesions (which may be melanoma), melanoma, or a history of melanoma
11. Any other conditions that, in the opinion of the investigator, would interfere with the evaluation of the results or constitute a health hazard for the patient
12. Allergic response to PPX or the inactive ingredients in its tablet formulation
13. Had previous treatment with dopamine agonists other than PPX within 14 days prior to the baseline visit
14. Had any other medical treatment for RLS besides the study medication within 14 days prior to the baseline visit
15. Had withdrawal symptoms of any medication at screening or at the baseline visit

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open label, single dose pharmacokinetic study in pediatric patients with a diagnosis of idiopathic Restless Legs Syndrome(RLS). For the dose MIRAPEX(0.5 mg),Only 2 subjects (12 to<18 years) were recruited and it was not likely that patients for this dose will be fully recruited so the recruitment was stopped and terminated for this dose only.
Groups:
- PPX (MIRAPEX®, 0.125 mg): Orally administered single daily maintenance dose of MIRAPEX® (0.125 mg) tablet per day in evening with 240 mL of water in a fasting state.
- PPX (MIRAPEX®, 0.25 mg): Orally administered single daily maintenance dose of MIRAPEX® (0.25 mg) tablet per day in evening with 240 mL of water in a fasting state.
- PPX (MIRAPEX®, 0.5 mg): Orally administered single daily maintenance dose of MIRAPEX® (0.5 mg) tablet per day in evening with 240 mL of water in a fasting state.
Period: Overall Study
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Started | 9 | 15 | 2
Completed | 9 | 14 | 1
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: The safety population comprised all patients who provided informed consent and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg) | Total
Number analyzed (Participants) | 9 | 15 | 2 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (4.3) | 11.4 (3.4) | 15.0 (0.0) | 11.4 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 2 | 12
  Male | 4 | 10 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Cmax,ss
Description: Maximum concentration of the Pramipexole (PPX) in plasma at steady state over a uniform dosing interval (Cmax,ss).
Time Frame: 0.25h before the drug administration on day1 and 0.5 h, 1 h, 2 h, 3 h, 5 h, 7h, 12h and 24h after the last drug administration on day 1.
Population: Pharmacokinetic Set (PK): All evaluable patients who received at least one dose of Pramipexole (PPX) between 0.125 and 0.5 mg were included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
ng/mL
  6 to <12 years (N=5, 9, 0) | 0.633 (26.2) | 1.13 (35.3) | NA (NA) — No patients were recruited for this category.
  12 to <18 years(N=4, 6, 2)) | 0.396 (30.0) | 0.677 (40.3) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the geometric mean (gMean) and geometric coefficient of variation (gCV) is not calculated according to internal rules.

2. Primary Outcome: Cmin,ss
Description: Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval (Cmin,ss).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
ng/mL
  6 to <12 years (N=5, 9, 0) | 0.0872 (35.5) | 0.136 (99.5) | NA (NA) — No patients were recruited for this category.
  12 to <18 years(N=4, 6, 2) | 0.0972 (37.5) | 0.122 (53.8) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

3. Primary Outcome: Cpre,N
Description: Predose concentration of the analyte in plasma at steady state immediately before administration of the next dose N (Cpre,N).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
ng/mL
  6 to <12 years (N=4, 8, 0) | 0.074 (17.3) | 0.147 (75.3) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=1, 5, 1) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | 0.112 (60.7) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

4. Primary Outcome: Cavg
Description: Average concentration of the analyte in plasma at steady state (Cavg).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
ng/mL
  6 to <12 years (N=5, 8, 0) | 0.213 (27.4) | 0.458 (42.8) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 0.137 (21.3) | 0.309 (35.2) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

5. Primary Outcome: Tmax,ss
Description: Time from dosing to maximum concentration at steady state (Tmax,ss).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
hours
  6 to <12 years (N=5, 9, 0) | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 3.00] | NA [NA to NA] — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 2) | 2.00 [0.50 to 2.00] | 1.96 [0.50 to 5.00] | NA [NA to NA] — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the median and range are not calculated according to internal rules.

6. Primary Outcome: Tmin,ss
Description: Time from dosing to minimum concentration at steady state (Tmin,ss ).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PK): All evaluable subjects who received at least one dose of Pramipexole (PPX) between 0.125 and 0.5 mg were included in the PK analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
hours
  6 to <12 years (N=5, 9, 0) | 12.0 [0.50 to 24.0] | 24.0 [0.25 to 24.0] | NA [NA to NA] — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 2) | 6.25 [0.50 to 12.0] | 23.9 [0.50 to 24.0] | NA [NA to NA] — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the median and range are not calculated according to internal rules.

7. Primary Outcome: AUCτ,ss
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval (AUCτ,ss ).
Time Frame: 0.25h before the drug administration on day 1 and 0.5 h, 1 h, 2 h, 3 h, 5 h, 7h, 12h and 24h after the last drug administration on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
ng*h/mL
  6 to <12 years (N=5, 8, 0) | 5.12 (27.4) | 11.0 (42.8) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 3.28 (21.3) | 7.42 (35.2) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

8. Primary Outcome: λz,ss
Description: Terminal rate constant in plasma at steady state (λz,ss ).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
1/h
  6 to <12 years (N=5, 8, 0) | 0.132 (22.6) | 0.107 (20.1) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 0.113 (1.88) | 0.0938 (25.4) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

9. Primary Outcome: t1/2,ss
Description: Terminal half-life of the analyte in plasma at steady state (t1/2,ss ).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
hours
  6 to <12 years (N=5, 8, 0) | 5.26 (22.6) | 6.50 (20.1) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 6.13 (1.88) | 7.39 (25.4) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

10. Primary Outcome: MRTpo,ss
Description: Mean residence time of the analyte in the body at steady state (MRTpo,ss).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
h
  6 to <12 years (N=5, 8, 0) | 8.19 (13.1) | 10.1 (19.5) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 9.47 (5.30) | 11.6 (23.3) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

11. Primary Outcome: CL/F,ss
Description: Apparent clearance of the analyte in the plasma after extravascular administration at steady state; F = absolute bioavailability factor (CL/F,ss ).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
mL/min
  6 to <12 years (N=5, 8, 0) | 284 (27.4) | 265 (42.8) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 444 (21.3) | 393 (35.2) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

12. Primary Outcome: Vz/F,ss
Description: Apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state (Vz/F,ss ).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
L
  6 to <12 years (N=5, 8, 0) | 129 (12.3) | 149 (29.7) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=4, 6,1) | 236 (19.4) | 251 (37.3) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

13. Primary Outcome: Ae 0-12,ss
Description: Amount of analyte that is eliminated in urine at steady state over a time interval t1to t2 (0-12h).
Time Frame: 12 hours after last study drug administration on day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
ng
  6 to <12 years (N=4, 6, 0) | 50600 (14.6) | 123000 (50.7) | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=3, 6, 0) | 55200 (41.5) | 82300 (52.7) | NA (NA) — No data was available of any patients for this category, so there was no data to analyse.

14. Primary Outcome: fe 0-12,ss
Description: Fraction of administered drug excreted unchanged in urine at steady state over a time interval t1 to t2 (fe 0-12,ss ).
Time Frame: 12 hours after last study drug administration on day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of PPX excreted
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
% of PPX excreted
  6 to <12 years (N=4, 2, 0) | 58.0 (14.6) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | NA (NA) — No patients were recruited for this category.
  12 to <18 years (N=2, 5, 0) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | 42.0 (48.1) | NA (NA) — No data was available of any patients for this category, so there was no data to analyse.

15. Primary Outcome: CLR,ss
Description: Renal clearance of the analyte at steady state (CLR(0-12),ss ).
Time Frame: 12h after last study drug administration on day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
mL/min
  6 to <12 years (N=4, 2, 0) | 201 (34.1) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | NA (NA) — No subjects were recruited for this category.
  12 to <18 years (N=2, 5, 0) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | 253 (34.1) | NA (NA) — No data was available of any patients for this category, so there was no data to analyse.

16. Primary Outcome: PTF
Description: Peak-trough fluctuation (PTF) is defined as the difference between Cmax and Cmin divided by Cavg and multiplied with 100% at steady-state.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of PTF
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
% of PTF
  6 to <12 years (N=5, 8, 0) | 250 (10.1) | 209 (31.8) | NA (NA) — No subjects were recruited for this category.
  12 to <18 years (N=4, 6, 1) | 216 (24.0) | 168 (34.2) | NA (NA) — The reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

17. Secondary Outcome: Number of Patients With Drug Related Adverse Events
Description: Number of patients with adverse events due to study drug.
Time Frame: From first drug administration until 24 hours after last study drug administration, upto 48 days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
participants | 1 | 0 | 1

18. Secondary Outcome: Vital Signs (Systolic and Diastolic Blood Pressure)
Description: Vital signs (Systolic and diastolic blood pressure (both supine and after standing for 1 minute)).
Time Frame: -0:15h(hours) pre-dose, and 0:30h, 1:00h, 2:00h, 3:00h, 5:00h, 7:00h, 12:00h, 24:00h post-dose.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
mmHg
  Systolic blood pressure-supine(N= 9,15,2): -0:15h | 109.33 (6.76) | 109.20 (10.80) | 117.00 (4.24)
  Systolic blood pressure-supine(N= 9,15,2): 0:30h | 112.89 (13.90) | 110.33 (14.07) | 116.00 (4.24)
  Systolic blood pressure-supine(N= 9,15,2): 1:00h | 113.00 (11.07) | 108.07 (12.92) | 105.50 (0.71)
  Systolic blood pressure-supine(N= 9,15,2): 2:00h | 111.00 (7.43) | 111.93 (13.79) | 113.00 (9.90)
  Systolic blood pressure-supine(N= 9,15,1): 3:00h | 106.89 (10.40) | 110.53 (11.34) | 113.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-supine(N= 9,15,1): 5:00h | 105.11 (12.71) | 108.80 (14.89) | 104.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-supine(N= 9,14,1): 7:00h | 108.44 (12.27) | 109.86 (14.11) | 108.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-supine(N= 9,14,1): 12:00h | 107.56 (16.38) | 106.93 (16.28) | 109.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-supine(N= 9,14,1): 24:00h | 109.22 (11.38) | 112.21 (13.76) | 120.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-supine(N= 9,15,2): -0:15 | 66.67 (7.35) | 65.73 (10.19) | 76.00 (0.00)
  Diastolic blood pressure-supine(N= 9,15,2): 0:30 | 68.67 (8.93) | 65.80 (12.62) | 73.00 (2.83)
  Diastolic blood pressure-supine(N= 9,15,2): 1:00 | 69.33 (6.52) | 65.73 (7.80) | 64.00 (12.73)
  Diastolic blood pressure-supine(N= 9,15,2): 2:00 | 66.00 (8.23) | 65.80 (8.76) | 75.00 (8.49)
  Diastolic blood pressure-supine(N= 9,15,1): 3:00 | 66.78 (9.36) | 65.40 (9.96) | 75.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-supine(N= 9,15,1): 5:00 | 64.22 (9.83) | 63.87 (9.78) | 70.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-supine(N= 9,14,1): 7:00 | 67.56 (13.47) | 62.43 (8.08) | 67.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-supine(N= 9,14,1): 12:00 | 70.00 (12.03) | 61.00 (9.12) | 66.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-supine(N= 9,14,1): 24:00 | 66.56 (6.00) | 65.71 (7.61) | 78.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-standing(N= 9,15,2):-0:15h | 109.89 (8.57) | 113.93 (9.97) | 122.00 (9.90)
  Systolic blood pressure-standing(N= 9,15,2): 0:30h | 113.56 (13.62) | 113.67 (13.69) | 115.50 (6.36)
  Systolic blood pressure-standing(N= 9,15,2): 1:00h | 110.11 (13.81) | 110.07 (14.26) | 125.50 (23.33)
  Systolic blood pressure-standing(N= 9,15,2): 2:00h | 110.33 (8.76) | 112.27 (12.26) | 115.00 (2.83)
  Systolic blood pressure-standing(N= 9,15,1): 3:00h | 110.11 (16.50) | 113.07 (16.15) | 108.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-standing(N= 9,14,1): 5:00h | 110.22 (11.88) | 111.93 (14.91) | 115.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-standing(N= 9,13,1): 7:00h | 109.11 (11.76) | 103.85 (17.56) | 65.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-standing(N=9,14,1): 12:00h | 108.22 (9.59) | 107.14 (15.83) | 100.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Systolic blood pressure-standing(N=9,14,1): 24:00h | 113.89 (11.25) | 115.50 (14.43) | 102.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolicblood pressure-standing(N=9,15,2): -0:15h | 68.11 (11.87) | 71.20 (8.09) | 86.00 (0.00)
  Diastolic blood pressure-standing(N=9,15,2): 0:30h | 70.11 (7.44) | 69.20 (12.11) | 80.00 (1.41)
  Diastolic blood pressure-standing(N=9,15,2): 1:00h | 69.22 (6.36) | 72.00 (9.54) | 91.00 (7.07)
  Diastolic blood pressure-standing(N=9,15,2): 2:00h | 71.11 (8.82) | 73.13 (9.36) | 86.50 (3.54)
  Diastolic blood pressure-standing(N=9,15,1): 3:00h | 72.67 (5.94) | 71.47 (8.98) | 79.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-standing(N=9,14,1): 5:00h | 74.00 (10.82) | 70.57 (9.20) | 98.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-standing(N=9,13,1):7:00h | 72.00 (13.01) | 66.69 (10.90) | 48.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolic blood pressure-standing(N=9,14,1):12:00h | 74.33 (11.19) | 70.07 (10.51) | 62.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Diastolicblood pressure-standing(N=9,14,1):24:00h | 73.11 (8.13) | 73.57 (9.62) | 84.00 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.

19. Secondary Outcome: Vital Signs (Pulse Rate)
Description: Vital signs (Pulse rate (both supine and after standing for 1 minute)).
Time Frame: -0:15h(hours) pre-dose, and 0:30h, 1:00h, 2:00h, 3:00h, 5:00h, 7:00h, 12:00h, 24:00h
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | PPX (MIRAPEX®, 0.125 mg) | PPX (MIRAPEX®, 0.25 mg) | PPX (MIRAPEX®, 0.5 mg)
Number analyzed (Participants) | 9 | 15 | 2
bpm
  Pulse rate-supine(N=9,15,2): -0:15h | 82.4 (18.6) | 73.3 (6.8) | 75.5 (24.7)
  Pulse rate-supine(N=9,15,2): 0:30h | 76.7 (17.5) | 78.0 (11.7) | 92.0 (32.5)
  Pulse rate-supine(N=9,15,2): 1:00h | 82.7 (22.2) | 75.2 (6.8) | 87.0 (36.8)
  Pulse rate-supine(N=9,15,2): 2:00h | 85.4 (19.6) | 77.9 (8.0) | 94.5 (26.2)
  Pulse rate-supine(N=9,15,1): 3:00h | 89.3 (19.1) | 79.9 (13.6) | 72.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate-supine(N=9,15,1): 5:00h | 82.7 (16.0) | 75.9 (6.9) | 77.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate-supine(N=9,14,1): 7:00h | 88.1 (18.1) | 72.0 (9.0) | 78.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate-supine(N=9,14,1): 12:00h | 77.8 (15.2) | 68.6 (6.2) | 69.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate-supine(N=9,14,1): 24:00h | 77.9 (13.6) | 77.6 (8.5) | 77.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate- standing(N=9,15,2):-0:15h | 90.8 (18.3) | 79.4 (8.7) | 99.0 (22.6)
  Pulse rate- standing(N=9,15,2): 0:30h | 84.7 (15.5) | 81.5 (12.2) | 103 (27.6)
  Pulse rate- standing(N=9,15,2): 1:00h | 94.8 (20.3) | 85.4 (10.9) | 123 (43.1)
  Pulse rate- standing (N=9,15,2): 2:00h | 92.8 (17.0) | 89.3 (11.2) | 121 (1.4)
  Pulse rate- standing (N=9,15,1): 3:00h | 99.0 (18.2) | 92.7 (12.9) | 109 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate- standing (N=9,14,1): 5:00h | 99.3 (27.0) | 87.1 (11.4) | 76.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate- standing (N=9,13,1): 7:00h | 100 (17.0) | 82.1 (14.4) | 72.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate- standing (N=9,14,1): 12:00h | 97.8 (12.4) | 81.2 (12.3) | 86.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.
  Pulse rate- standing (N=9,14,1): 24:00h | 90.0 (18.8) | 85.8 (6.7) | 86.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable.

ADVERSE EVENTS:
Time Frame: From first drug administration until 24 hours after last study drug administration, upto 48 days
Groups:
- MIRAPEX® (0.125 mg): Orally administered single daily maintenance dose of MIRAPEX® (0.125 mg) tablet per day in evening with 240 mL of water in a fasting state.
- MIRAPEX® (0.25 mg): Orally administered single daily maintenance dose of MIRAPEX® (0.25 mg) tablet per day in evening with 240 mL of water in a fasting state.
- MIRAPEX® (0.5 mg): Orally administered single daily maintenance dose of MIRAPEX® (0.5 mg) tablet per day in evening with 240 mL of water in a fasting state.
Arm/Group | MIRAPEX® (0.125 mg) | MIRAPEX® (0.25 mg) | MIRAPEX® (0.5 mg)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/15 | 0/2
Other Adverse Events (participants affected / at risk) | 2/9 | 3/15 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIRAPEX® (0.125 mg) (N=9) | MIRAPEX® (0.25 mg) (N=15) | MIRAPEX® (0.5 mg) (N=2)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 1 | 0
Infusion site irritation (General disorders) | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 1 | 0
Vessel puncture site erythema (General disorders) | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.